CLINICAL TRIAL: NCT04826796
Title: Feasibility and Effectiveness of WhatsApp Online Group on Breastfeeding by Peer Counsellors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BFPSW
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Breastfeeding, Exclusive; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whatsapp intervention group (Experimental): In addition to standard care, participants will be included into a peer support Whatsapp group on Whatsapp with other participants and trained peer supporters after study entry. Standard weekly prompt text messages will be sent to the group by peer supporters to encourage questions and discussion related to breastfeeding. Peer supporters will provide breastfeeding and emotional support. Intervention will last for 6 months after birth.
  Interventions: Behavioral: WhatsApp peer support
- Control group (No Intervention): Participants in the control group will continue to receive standard care.

INTERVENTIONS:
Behavioral: WhatsApp peer support — Trained peer supporters will provide breastfeeding and emotional support for participants in the WhatsApp group.
  Arms: Whatsapp intervention group

SUMMARY:
Due the uncertainty of the pandemic wave and government restrictions that may affect health care services and behaviour, alternative mhealth strategies should be explored to identify breastfeeding support or problems early to prevent subsequent cessation that may affect mother and child health. It is also important to understand the feasibility of a WhatsApp online group on breastfeeding by peer counsellors during postnatal period and the acceptability of such intervention. Therefore this study will provide preliminary information necessary for implementation of a full RCT of mhealth intervention in the future. The aim of this study is to examine the feasibility and effectiveness of a WhatsApp online peer support group program in improving breastfeeding practices.

There have been no published studies that have examined the feasibility and acceptability of a Whatsapp online group on breastfeeding for postnatal women in Hong Kong. Given the significant pandemic problem that may affect health services and health behavior of pregnant women, the proposed study will contribute substantial new information about the feasibility and potential implications for future care pathways for postnatal women. Such information will be invaluable to public health professional working to breastfeeding promotion and to health policy makers in setting institutional policies.

DETAILED DESCRIPTION:
Mobile health (mhealth) refers to delivering health care and health promotion through mobile devices [1]. Advances of mobile technologies have led to increased use of mhealth interventions for effective healthy infant feeding practices and breastfeeding promotion. A meta-analysis reviewed that mhealth significantly improved exclusive breastfeeding initiation, breastfeeding attitude and knowledge [2]. Whether more interactive and adaptive mHealth platforms, including smartphone apps and social networking tools, could further improve breastfeeding outcomes remains understudied. Smartphones have become new channels and tools for information acquisition and exchange and have been well adopted by the general public. In 2019, the number of smartphone users in Hong Kong was estimated to reach 6.5 million. By the year 2025, it is predicted that 93% of the population in Hong Kong will use a smartphone [3]. Among instant messaging apps for smartphones, WhatsApp is regarded as one of the largest social network platforms used in Hong Kong. WhatsApp is a free all in one communications app widely used for sending text and voice messages, video calls. Online discussion platforms have been used, acceptable, affordable and accessible in previous years for promoting physical activity [4], a healthy diet [5], smoking cessation [6] and reducing alcohol use [7]. Interventions using these communication tools tend to have high uptake due to personalized intervention and instant response without having time and location limitations. Whether WhatsApp can be used as a communication tool to positively change selected behaviours has yet to be assessed its effects on breastfeeding outcomes.

With the current pandemic and social distancing measures, this study offers insight on the practicality and feasibility of supporting Chinese mothers who are housebound due to Chinese traditional cultural "doing the month" in which Chinese mothers are housebound during the first month post-birth. In addition, due to the pandemic, there is limited face to face antenatal and postnatal support from the health services. Unresolved problems and inadequate support with infant feeding may result in a decision to stop exclusively breastfeeding. Our previous qualitative study suggested that WhatsApp messaging might be a viable way of promoting breastfeeding (unpublished data). Therefore, a pilot study is developed to address an important service gap in Hong Kong to promote and sustain exclusive breastfeeding. However, there might be potential barriers to successful implementation and to evaluating the effectiveness of the innovation intervention. This is the first WhatsApp breastfeeding support programme provided by peer supporters in Hong Kong. In Hong Kong, the most recent breastfeeding survey showed that the exclusive breastfeeding rate at 6 months was 26.3% in Hong Kong [8]. Furthermore, more than 88% of mothers initiated breastfeeding but half of breastfeeding mothers never exclusively breastfed their babies [8]. Despite the importance of exclusive breastfeeding for the first 6 months postpartum, the maintenance of exclusive breastfeeding is a major public health issue particularly in Hong Kong where the rate on exclusive breastfeeding duration indicated that it tailed off during the first 2 months [8]. This indicates novel approaches are needed to engage hard to reach mothers who encounter breastfeeding problems or support during the first 6 months.

Existing services mainly target mothers in clinical or primary care settings delivered by health professionals for promoting breastfeeding. Hong Kong has an extensive smartphone penetration rate (78% in 2020). Therefore, before proceeding with a full scale randomized controlled trial (RCT), a feasibility and pilot study is needed to identify if a WhatsApp online group on breastfeeding by peer counsellors, delivered through instant/video messaging support, designed to improve breastfeeding outcomes is feasible and acceptable. The main objective of the study is to determine the feasibility of conducting a WhatsApp online group on breastfeeding by peer counsellors over a six-month period in postpartum Chinese women in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Primiparous
* Intend to breastfeed
* had a singleton pregnancy
* had term infant (37-42 weeks gestation)
* Cantonese speakers
* Hong Kong residents
* had no serious medical or obstetrical complications

Exclusion Criteria:

* Infant is <37 weeks gestation
* Infant has an Apgar score <8 at five minutes
* Infant has a birthweight <2500 grams
* Infant has any severe medical conditions or congenital malformations
* Infant is placed in the special care baby unit for more than 48 hours after birth
* Infant is placed in the neonatal intensive care unit at any time after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants are included
Enrollment: 43 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in proportion of participants who are exclusively breastfeeding | At 1, 2, 4, and 6 months postpartum
  The number of participants who are exclusively breastfeeding at each time point.
Change in proportion of participants who are any breastfeeding | At 1, 2, 4, and 6 months postpartum
  The number of participants who are any breastfeeding at each time point.

SECONDARY OUTCOMES:
Breastfeeding self-efficacy | At baseline and 2 month postpartum
  Breastfeeding efficacy measured using Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF). BSES-SF is a 14-item scale with total score ranging from 14 to 70. A higher score indicates higher breastfeeding self-efficacy.
Breastfeeding attitude | At baseline and 2 month postpartum
  Attitude towards breastfeeding measured using the Iowa Infant Feeding Attitude Scale (IIFAS). IIFAS is a 17-item scale with total score ranging from 17 to 85. A higher score indicates a more favourable attitude towards breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Lok, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Premji S. Mobile health in maternal and newborn care: fuzzy logic. Int J Environ Res Public Health. 2014 Jun;11(6):6494-503. doi: 10.3390/ijerph110606494. PMID 25003177
- [Background] Lau Y, Htun TP, Tam WS, Klainin-Yobas P. Efficacy of e-technologies in improving breastfeeding outcomes among perinatal women: a meta-analysis. Matern Child Nutr. 2016 Jul;12(3):381-401. doi: 10.1111/mcn.12202. Epub 2015 Jul 21. PMID 26194599
- [Background] Statista. Available from: www.statista.com Access date 20-11-2020
- [Background] Rovniak LS, Kong L, Hovell MF, Ding D, Sallis JF, Ray CA, Kraschnewski JL, Matthews SA, Kiser E, Chinchilli VM, George DR, Sciamanna CN. Engineering Online and In-Person Social Networks for Physical Activity: A Randomized Trial. Ann Behav Med. 2016 Dec;50(6):885-897. doi: 10.1007/s12160-016-9814-8. PMID 27405724
- [Background] Ahmad N, Shariff ZM, Mukhtar F, Lye MS. Family-based intervention using face-to-face sessions and social media to improve Malay primary school children's adiposity: a randomized controlled field trial of the Malaysian REDUCE programme. Nutr J. 2018 Aug 2;17(1):74. doi: 10.1186/s12937-018-0379-1. PMID 30071855
- [Background] Cheung YTD, Chan CHH, Ho KS, Fok WP, Conway M, Wong CKH, Li WHC, Wang MP, Lam TH. Effectiveness of WhatsApp online group discussion for smoking relapse prevention: protocol for a pragmatic randomized controlled trial. Addiction. 2020 Sep;115(9):1777-1785. doi: 10.1111/add.15027. Epub 2020 Mar 20. PMID 32107817
- [Background] Byrnes HF, Miller BA, Grube JW, Bourdeau B, Buller DB, Wang-Schweig M, Woodall WG. Prevention of alcohol use in older teens: A randomized trial of an online family prevention program. Psychol Addict Behav. 2019 Feb;33(1):1-14. doi: 10.1037/adb0000442. Epub 2019 Jan 14. PMID 30640504
- [Background] Department of Health. Breastfeeding Survey 2019. Available from: https://www.fhs.gov.hk/english/archive/files/reports/BF_survey_2019.pdf.
- [Derived] Fan HSL, Ho MY, Ko RWT, Kwok JYY, Chau PH, Wong JYH, Wang MP, Lok KYW. Feasibility and effectiveness of WhatsApp online group on breastfeeding by peer counsellors: a single-blinded, open-label pilot randomized controlled study. Int Breastfeed J. 2022 Dec 22;17(1):91. doi: 10.1186/s13006-022-00535-z. PMID 36544208
- [Derived] Lok KY, Ko RW, Fan HS, Chau PH, Wong JY, Wang MP, Tsang V. Feasibility and Acceptability of an Online WhatsApp Support Group on Breastfeeding: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Mar 9;11(3):e32338. doi: 10.2196/32338. PMID 35262504